CLINICAL TRIAL: NCT04575233
Title: Laparoscopic- Vs Ultrasound-guided Transversus Abdominis Plane Block in Laparoscopic Colectomy: a Prospective Randomized Controlled Trial
Brief Title: A Study to Compare Laparoscopic to Echographic Assisted Transversus Abdominis Plane Block in Laparoscopic Colectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Davide La Regina (Other)
Responsible Party: Sponsor-Investigator, Davide La Regina, Principal Investigator, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAP block
Record Dates: First submitted 2020-09-18; First posted 2020-10-05 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Laparoscopic Colectomy; Pain, Postoperative
Keywords: Transversus Abdominis Plane (TAP) Block; Local Anesthetic Infiltrations
MeSH Terms: conditions — Pain, Postoperative; Bites and Stings | interventions — Dental Occlusion; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Transversus Abdominis Plane (L-TAP) group (Experimental): Patients will undergo the planned laparoscopic colectomy according to the standard of treatment. A solution of 15 ml of Ropivacaine (0.2%) is then injected for postoperative pain under laparoscopic control
  Interventions: Procedure: laparoscopic-assisted Transversus Abdominis Plane (TAP) block; Drug: Ropivacaine
- Ultrasound Transversus Abdominis Plane (U-TAP) group (Active Comparator): Patients will undergo the planned laparoscopic colectomy according to the standard of treatment. A solution of 15 ml of Ropivacaine (0.2%) is then injected for postoperative pain under ultrasound control
  Interventions: Procedure: ultrasound-assisted Transversus Abdominis Plane (TAP) block; Drug: Ropivacaine

INTERVENTIONS:
Procedure: laparoscopic-assisted Transversus Abdominis Plane (TAP) block — The anterior axillary line is used as landmarks. After insertion of the optic trocar, the peritoneum is visualized. A 14 Gauge needle is inserted 2 cm cranially respect the taken landmark through the skin until the penetration of the internal and external oblique fascias, identified as sudden lowering of resistance. A solution of 15 ml of Ropivacaine (0.2%) is then injected. The procedure is performed then 2 cm caudal to the first landmark on the same side.
  The procedure is than repeated identically on the contralateral side.
  Arms: Laparoscopic Transversus Abdominis Plane (L-TAP) group
Procedure: ultrasound-assisted Transversus Abdominis Plane (TAP) block — Whilst the patient is in the supine position, a high frequency ultrasound probe is placed transverse to the abdominal wall between the costal margin and iliac crest. The needle is introduced in plane of the ultrasound probe directly under the probe and advanced until it reaches the plane between the internal oblique and transversus abdominis muscles. Then 15 ml of local anaesthetic solution is injected. The needle is than retracted until its tip is positioned in the fascial plane between the internal and the external oblique muscles and a second bolus of 15 ml of local anaesthetic is injected. The procedure is than repeated identically on the contralateral side.
  Arms: Ultrasound Transversus Abdominis Plane (U-TAP) group
Drug: Ropivacaine — a solution of 15 ml of Ropivacaine (0.2%) is injected for the treatment of post-operative pain after minimally invasive surgery (TAP block)

SUMMARY:
The purpose of this study is to compare the postoperative pain, the time needed and other clinical outcomes in patients who, during laparoscopic colectomy, will be injected with a local anesthetic (Ropivacaine) through an ultrasound guided technique performed by the anaesthesiologist or throught a laparoscopic assisted technique performed by the surgeon

ELIGIBILITY:
Inclusion Criteria:

* Patients candidates to laparoscopic colorectal surgery
* Signed informed consent

Exclusion Criteria:

* Age < 18 years old
* Pregnancy
* Allergy to local anaesthetics
* Spinal or epidural analgesia
* Acute inflammatory abdominal pathologies
* Chronic pain syndrome
* Contraindications to nonsteroidal anti-inflammatory drugs (NSAIDS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Opioids consumption | 24 hours from surgery
  Opioid consumption measured in morphine milligram equivalents (MME) per day

SECONDARY OUTCOMES:
Opioid consumption within the first 48 hours after the operation | 48 hours from surgery
  Opioid consumption measured in morphine milligram equivalents (MME) per day
postoperative pain | at 3, 6, 12, 24 hours from surgery
  Postoperative pain on the visual analogue scale (VAS) at 3, 6, 12, 24 hours. This visual analogue scale measures the subjective pain: patients indicate a position along a continuous line between two end-points to specify their level of pain. Absence of pain is represented by 0 while 10 corresponds to the maximum of pain.
length of hospital stay | during hospitalization,approximately 6 days
  number of days the participant is being hospitalized
Time required to perform the (Transversus Abdominis Plane) TAP block | during procedure

CONTACTS AND LOCATIONS:
Overall Officials: Davide La Regina, MD, Study Chair — Ente Ospedaliero Cantonale (EOC)
Locations (2):
- Switzerland (2):
  - Ospedale Regionale Bellinzona e Valli, Ente Ospedaliero Cantonale, Bellinzona
  - Ospedale Regionale di Lugano, Civico e Italiano - Ente Ospedaliero Cantonale, Lugano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] La Regina D, Popeskou SG, Saporito A, Gaffuri P, Tasciotti E, Dossi R, Christoforidis D, Mongelli F. Laparoscopic versus ultrasound-guided transversus abdominis plane block in colorectal surgery: a non-inferiority, multicentric randomized double-blinded clinical trial. Colorectal Dis. 2023 Sep;25(9):1921-1928. doi: 10.1111/codi.16689. Epub 2023 Jul 31. PMID 37525414